CLINICAL TRIAL: NCT03283150
Title: Effects of Anesthesia Drugs on Neuronal Activity in the Basal Ganglia and Thalamus During Deep Brain Stimulation Electrode Implantation Surgery
Brief Title: Deep Brain Stimulation (DBS) Sedation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to a decrease in scheduled study-eligible patients, we terminated the study prematurely
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2016-1420; A530900 (Other: UW Madison); SMPH\ANESTHESIOLOGY\ANESTHESIO (Other: UW Madison); Protocol Version 2/17/2020 (Other: UW Madison)
Record Dates: First submitted 2017-09-06; First posted 2017-09-14 (Actual); Results first posted 2023-03-27 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Brain; Sedation
Keywords: Deep Brain Stimulation(DBS); Sedation; DBS Implantation; Microelectrode recording(MER)
MeSH Terms: interventions — Remifentanil; Propofol; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Remifentanil (Active Comparator): Remifentanil will be administered to subjects during microelectrode recordings (MER).
  Interventions: Drug: Remifentanil
- Propofol (Active Comparator): Propofol will be administered to subjects during MER.
  Interventions: Drug: Propofol
- Dexmedetomidine (Active Comparator): Dexmedetomidine will be administered to subjects during MER.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Remifentanil — Remifentanyl will be administered for 10 -15 minutes before initiating the MER phase and the patient will be allow to wake up and the bispectral index (BIS) values to normalize to awake level for the MER.
  Arms: Remifentanil
Drug: Propofol — Propofol will be administered for 10 -15 minutes before initiating the MER phase and the patient will be allow to wake up and the BIS values to normalize to awake level for the MER.
  Arms: Propofol
Drug: Dexmedetomidine — Dexmedetomidine will be administered for 10 -15 minutes before initiating the MER phase and the patient will be allow to wake up and the BIS values to normalize to awake level for the MER.
  Arms: Dexmedetomidine

SUMMARY:
Deep brain stimulation (DBS) of different brain nuclei is a treatment for multiple brain disorders. The subthalamic nucleus (STN) and globus pallidus have been used to treat advanced Parkinson's disease for a long time. The ventral intermediate nucleus of the thalamus is an effective target for treating essential tremor patients. STN and the internal segment of the globus pallidus are useful targets for treating dystonia.

To achieve this optimal electrode localization, many centers perform electrophysiological mapping of the target nuclei using microelectrode recording (MER). This way they can achieve precise localization of the electrode. During the mapping procedure, microelectrodes are passed through the target nuclei, and the electrical neuronal activity is observed and recorded. The surgical team can identify the precise location of the target nuclei and its borders according to the typical activity of its neurons.

This study will compare the activity of neurons in several DBS targets before, during and after sedation with propofol, remifentanil and dexmedetomidine. The goal is to understand the effects of anesthetics on the neuronal activity in these targets, allowing us to choose the most appropriate sedation protocol to use during implantation of DBS electrodes in deep brain structures (bearing in mind that each structure may have a different optimal protocol).

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) of different brain nuclei is evolving as an essential component of the treatment for multiple brain disorders. The subthalamic nucleus (STN) and globus pallidus have been used to treat advanced Parkinson's disease for a long time. The ventral intermediate nucleus of the thalamus is an effective target for treating essential tremor patients. STN and the internal segment of the globus pallidus are useful targets for treating dystonia. Aside from movement disorders DBS has demonstrated efficacy in the treatment of other conditions such as chronic pain, obsessive compulsive disorder, depression and epilepsy. For these illnesses the specific brain region targeted depends upon the illness and the patient's characteristics. As the indications for DBS increase in number, so grows the number of patients that may be helped by this treatment. Increasing numbers of patients are undergoing these procedures for various maladies at our center and at other locations throughout the nation.

To achieve optimal clinical results and avoid side effects, the DBS electrode has to be implanted precisely within the targeted region. This was demonstrated elegantly for parkinsonian patients and the dorsolateral STN, but is likely to be the case for most DBS indications. To achieve this optimal electrode localization, many centers perform electrophysiological mapping of the target nuclei using microelectrode recording (MER). This way they can achieve precise localization of the electrode. During the mapping procedure, microelectrodes are passed through the target nuclei, and the electrical neuronal activity is observed and recorded. The surgical team can identify the precise location of the target nuclei and its borders according to the typical activity of its neurons.

Dexmedetomidine, propofol and remifentanyl are often used in awake neurosurgical procedures. Dexmedetomidine provides sedation and amnesia with minimal respiratory depression, and improves perioperative hemodynamic stability in neurosurgical patients. Propofol and remifentanil have a much shorter duration of action, and thus allow rapid titration. Both these agents allow reliable and safe sedation for awake craniotomies. However, the effects of any of these three agents on the electrical activity, and whether they will allow safe sedation during DBS electrode implantation at different targets and in different clinical conditions is unclear.

This study will compare the activity of neurons in several DBS targets before, during and after sedation with propofol, remifentanil and dexmedetomidine. The goal is to understand the effects of anesthetics on the neuronal activity in these targets, allowing the study team to choose the most appropriate sedation protocol to use during implantation of DBS electrodes in deep brain structures (bearing in mind that each structure may have a different optimal protocol).

The primary aim is to document the effects of commonly used anesthetic drugs on the neuronal activity during MER in different brain structures that are used as targets for DBS implantation.

The secondary aims is to Identifying effective sedation regimens for the different DBS targets; (2) Documenting the time course of the different drug's effect on the neuronal activity. Having this information will allow planning and performing sedation during the procedure prior to the MER without affecting the quality of the MER. This may prove useful in cases where no sedation regimen is completely devoid of effect on the MER; (3) Creating a database that includes the neuronal activity changes at multiple brain regions under the effect of different sedation drugs to enable further study of the effects of anesthetics on brain regions and the mechanisms underlying loss of consciousness.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled to undergo DBS electrode implantation surgery with MER that agree to participate in the experiment and sign an informed consent are candidates to participate in the study, unless one of the exclusion criteria is met

Exclusion Criteria:

1. Known or suspected obstructive sleep apnea.
2. Suspected difficult intubation.
3. Pregnancy (pregnancy test is standard care for women of childbearing age)
4. Under 18 years of age or over 85 years of age
5. Cognitive disability impairing understanding the experiment or signing the informed consent form.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey A Amlong, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Background] Raz A, Eimerl D, Zaidel A, Bergman H, Israel Z. Propofol decreases neuronal population spiking activity in the subthalamic nucleus of Parkinsonian patients. Anesth Analg. 2010 Nov;111(5):1285-9. doi: 10.1213/ANE.0b013e3181f565f2. Epub 2010 Sep 14. PMID 20841416

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Remifentanil | Propofol | Dexmedetomidine
Started | 20 | 0 | 0
Completed | 14 | 0 | 0
Not Completed | 6 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects were accrued to the baseline propofol and dexmedetomidine groups. The study was stopped early due to COVID decreasing participant flow and the frequency of the surgery dropping due to surgeon loss.
Groups:
- Remifentanil: Remifentanil will be administered to subjects during microelectrode recordings (MER).
  Remifentanil: Remifentanyl will be administered for 10 -15 minutes before initiating the MER phase and the patient will be allow to wake up and the BIS values to normalize to awake level for the MER.
- Total: Total of all reporting groups
Arm/Group | Remifentanil | Propofol | Dexmedetomidine | Total
Number analyzed (Participants) | 20 | 0 | 0 | 20
Age, Continuous [Mean (Full Range); unit: years] | 60 [52 to 67] |  |  | 60 [52 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 |  |  | 5
  Male | 15 |  |  | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  |  | 0
  Not Hispanic or Latino | 18 |  |  | 18
  Unknown or Not Reported | 2 |  |  | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 0 |  |  | 0
  White | 18 |  |  | 18
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 2 |  |  | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 |  |  | 20

OUTCOME MEASURES:

1. Primary Outcome: Sedatives Drugs Effects - Percent Change in Root Mean Square (RMS) of Electrical Activity
Description: Effects of propofol, remifentanil and dexmedetomidine on the neuronal activity during microelectrode recording (MER) in different brain structures that are used as target for DBS implantation will be measure.
  The RMS of the electrical activity as a measure of the spiking rate of neurons in the vicinity of the electrode tip. normalize the RMS to the baseline value recorded at the first 2-5 minutes of MER (before entering the target area) to compensate for differences between patients and recording electrodes. In order to calculate the change in the normalized RMS following sedation the investigators will compare the mean RMS during 2 minutes of the stable recording of the pre-sedation baseline to the mean RMS during stable sedation and following recovery.
Time Frame: 45 minutes
Population: No subjects were accrued into the propofol or dexmedetomidine groups as COVID-19 struck and the number of procedures performed decreased substantially during and post-COVID.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Remifentanil | Propofol | Dexmedetomidine
Number analyzed (Participants) | 14 | 0 | 0
percent change | 2.69 (0.37) |  |

2. Secondary Outcome: Mean Time in Minutes From Sedation to Recovery
Description: This outocme meadsures the mean time from sedation to recovery.
Time Frame: up to 57 minutes
Population: No subjects were accrued to the propofol or dexmedetomidine groups.
Measure: Mean (Full Range); unit: minutes
Arm/Group | Remifentanil | Propofol | Dexmedetomidine
Number analyzed (Participants) | 14 | 0 | 0
minutes | 29.43 [11 to 57] |  |

3. Secondary Outcome: Number of Individuals Examined for Neuronal Activity Changes at Multiple Brain Regions Under the Effect of Different Sedative Drugs
Description: The number of subjects examining the neuronal activity changes at multiple brain regions under the effect of different sedation drugs to enable further study of the effects of anesthetics on brain regions and the mechanisms underlying loss of consciousness.
Time Frame: 1hrs 30 min
Population: No subjects were accrued to the propofol or dexmedetomidine groups due to COVID and the decrease in the frequency of the surgery being performed at the hospital.
Measure: Count of Participants; unit: Participants
Arm/Group | Remifentanil | Propofol | Dexmedetomidine
Number analyzed (Participants) | 14 | 0 | 0
Participants | 14 | 0 | 0

ADVERSE EVENTS:
Time Frame: during 1 study visit, up to 4 hours
Description: Participants were only recruited into the Remifentanil arm. Study was terminated early per COVID-19 pandemic.
Arm/Group | Remifentanil | Propofol | Dexmedetomidine
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/14 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT03283150/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT03283150/ICF_001.pdf